CLINICAL TRIAL: NCT00718926
Title: The Evaluation of Thiol Redox Status in Conjunctiva of Dry Eye Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meiji University of Oriental Medicine (Other)
Collaborators: Kyoto Prefectural University of Medicine (Other)
Responsible Party: Jun Yamada MD. PhD., Meiji University of Oriental Medicine
Other Study IDs: C244
Record Dates: First submitted 2008-07-18; First posted 2008-07-21 (Estimated); Last update posted 2008-07-21 (Estimated); Status verified 2008-05

CONDITIONS: Dry Eye Disease
Keywords: dry eye; Thiol redox; Oxidative stress
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Control
Biospecimen Retention: Samples Without DNA — After application of anethesia eyedrops, nitrocel membrane is put ocular surface. Then, removed the membrane. This method is commonly used clinically.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Sjogren: Sjogren syndrome with dry eye
- non-Sjogren: dry eye without Sjogren syndrome
- Short-BUT: Dry eye by shortened tear break up time
- control: normal patients

SUMMARY:
Dry eye disease is related with oxidative stress at the ocular surface. GSH is one of the key factor of protect from oxidative stress. To evaluate thiol status of ocular surface cells by monitoring GSH concentration, we can evaluate the severity of dry eye.

DETAILED DESCRIPTION:
The conjunctival cells are collected by impression cytology. Those cells are stained with 100 mM of monochlorobimane (MCB, M-1381, Molecular Probes, Eugene, OR) and propidium iodide (PI). Fluorescent intensity, reflecting the amount of icGSH, was inspected under a confocal laser scan microscope. To detect the GSH levels we used a fluorescent MCB probe with excitation and emission wavelengths of 405 nm and 410-480 nm, respectively. The cell-permeating MCB probe is non-fluorescent but forms a fluorescent adduct with GSH in a reaction catalyzed by glutathione-S-transferase.

ELIGIBILITY:
Inclusion Criteria:

* dry eye patients
* control volunteers

Exclusion Criteria:

* Young (less than 20) patients
* The patients who rejected this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The dry eye patients at the clinic of Kyoto Prefectural University of Medicine hospital
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-08; Primary Completion 2008-12 (Estimated); Study Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Tear amount, tear break up time, and so on are measured clinically. The thiol redox status is measured by staining the membrane. | Once a month (totally 2-4 times) at the clinic

CONTACTS AND LOCATIONS:
Locations (1):
- Kyoto Prefectural University of Medicine hospital, Kyoto, Japan